CLINICAL TRIAL: NCT05412043
Title: Walking-related Fatigability in Persons With Multiple Sclerosis: Psychometric Properties of Cognitive and Coordination Fatigability Assessment & Proof-of-concept of a Rehabilitation Intervention
Brief Title: Fatigability in Persons With Multiple Sclerosis: Inputs From Cognition, Walking and Coordination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Revalidatie & MS Centrum Overpelt (Other); National MS Center Melsbroek (Other)
Responsible Party: Principal Investigator, Peter Feys, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Fatigability-MS-001
Record Dates: First submitted 2021-08-23; First posted 2022-06-09 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Walking-fatigability; cognitive-fatigability; coordination-fatigability; Psychometric properties
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dance Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Persons with MS - Dance group (Experimental): 12 pwMS in the Dance Therapy intervention
  Interventions: Behavioral: Dance therapy; Other: Psychometric properties (Validity, Reliability) of interlimb coordination- and cognitive-fatigability
- persons with MS - excercise group (Active Comparator): 12 pwMS in the exercise (placebo) group
  Interventions: Other: Psychometric properties (Validity, Reliability) of interlimb coordination- and cognitive-fatigability
- Healthy controls (Placebo Comparator)
  Interventions: Other: Psychometric properties (Validity, Reliability) of interlimb coordination- and cognitive-fatigability

INTERVENTIONS:
Behavioral: Dance therapy — The dance group will attend choreo-based dance therapy which includes both cognitive training to remember the choreo's and motor training to execute them (with and without music). Each session will consist of a ten-minute warm up, dance training and a ten-minute cool down. The participants will be taught three choreographies, which will increase in difficulty level. 1) floor work on a slow rhythm with focus on proprioception, abdominal muscle strength, coordination and working memory. 2) slow paced with a group part and a canon part with focus on working memory, static and dynamic balance and strength. Furthermore, it will require dynamic balance, walking and cognition. 3) higher rhythm and will be danced with a cane which will require more speed, coordination and dual tasking.
  Arms: Persons with MS - Dance group
Other: Psychometric properties (Validity, Reliability) of interlimb coordination- and cognitive-fatigability — The study consists of 2 test sessions, separated by 5-7 days of interval. The sessions 1 and 2 will be composed of cognitive test battery, questionnaires to be filled, information about the use of actigraph, clinical outcomes and interlimb coordination tests

SUMMARY:
Walking impairments occur in 93% of persons with MS (pwMS) within 10 years of diagnosis. Besides the impact of muscle weakness or hypertonia, one is increasingly aware about the symptom of fatigability. Motor and cognitive fatigability is a change in performance over time depending on the tasks and circumstances. It was shown that up to half of disabled pwMS slow down during walking, impacting on real life mobility. Walking function is related to functional muscle strength, balance and centrally mediated coordination deficits but also cognitive function. Preliminary data conducted by our research group has shown that people with MS with walking fatigability had a significant decrease in movement amplitude during a bipedal coordination task in sitting position. However, the psychometric properties such as within-session and test-retest reliability of bipedal function has not yet been determined. In addition, so far, no interventional research has included exclusively people with MS with walking-related fatigability. It is unknown if the downward curve in walking speed and coordination can be reversed by multi-model interventions.

The study will have two parts (A and B). Part A investigates psychometric properties of outcome measures related to fatigability in healthy controls, persons with MS with and without fatigability during walking. Part B is an intervention study in persons with MS and fatigability, comparing dance with a sham intervention, and its effects primarily on fatigability outcomes.

DETAILED DESCRIPTION:
The study will have two parts (A and B). Part A includes 60 persons with Multiple Sclerosis (pwMS) and 30 healthy controls. The study consists of 2 test sessions, separated by 5-7 days of interval. The sessions 1 and 2 will be composed of cognitive test battery, questionnaires to be filled, information about the use of actigraph, clinical outcomes and interlimb coordination tests.

In the Part B the investigators propose a pilot randomized controlled trial with dance therapy to improve fatigability in pwMS. The study includes 24 pwMS presenting walking fatigability. The participants will be randomly allocated by group (n=3-4), by a person independent from the research, into the intervention group (Dance Therapy) or the active control group (control exercise). Interventions take place in groups of 3 or 4 people with MS, twice a week for eight weeks, complementary to their usual care or conventional physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Persons with MS presenting walking-related fatigability (Distance walk index ≤-10);
* age between 30 and 70 years old;
* a diagnosis of MS (2017 revisions of the McDonalds criteria) with Expanded Disability Status Scale (EDSS) 4 up to 6.5.
* no relapses >1 month preceding the start of the study
* ability to walk for 6 minutes without rest.

Exclusion Criteria:

* Cognitive impairment hindering understanding of study instructions,
* pregnancy
* musculoskeletal disorders in the lower limbs not related to MS.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
The phase coordination index (PCI) | baselline
  The phase coordination index (PCI) will be used to analyse the consistency and accuracy in generating antiphase left-right knee movements on an instrumented chair. Participants will be instructed to perform antiphase movements of knee flexion and extension.
The phase coordination index (PCI) | Day 7
  The phase coordination index (PCI) will be used to analyse the consistency and accuracy in generating antiphase left-right knee movements on an instrumented chair. Participants will be instructed to perform antiphase movements of knee flexion and extension.
The phase coordination index (PCI) | week 8
  The phase coordination index (PCI) will be used to analyse the consistency and accuracy in generating antiphase left-right knee movements on an instrumented chair. Participants will be instructed to perform antiphase movements of knee flexion and extension.
Movement Amplitude- Chair Coordination test | Baseline
  Participants will be instructed to perform antiphase movements of knee flexion and extension on an instrumented chair. Intralimb spatiotemporal parameters per cycle of successive peak extension positions, and averaged per minute will include movement amplitude: peak-to-peak amplitude for each individual cycle.
Movement Amplitude- Chair Coordination test | Day 7
  Participants will be instructed to perform antiphase movements of knee flexion and extension on an instrumented chair. Intralimb spatiotemporal parameters per cycle of successive peak extension positions, and averaged per minute will include movement amplitude: peak-to-peak amplitude for each individual cycle.
Movement Amplitude- Chair Coordination test | Week 8
  Participants will be instructed to perform antiphase movements of knee flexion and extension on an instrumented chair. Intralimb spatiotemporal parameters per cycle of successive peak extension positions, and averaged per minute will include movement amplitude: peak-to-peak amplitude for each individual cycle.
Movement Frequency- Chair Coordination test | Baseline
  Participants will be instructed to perform antiphase movements of knee flexion and extension on an instrumented chair. Intralimb spatiotemporal parameters per cycle of successive peak extension positions, and averaged per minute will include movement frequency: the number of complete movements performed during one minute.
Movement Frequency- Chair Coordination test | Day 7
  Participants will be instructed to perform antiphase movements of knee flexion and extension on an instrumented chair. Intralimb spatiotemporal parameters per cycle of successive peak extension positions, and averaged per minute will include movement frequency: the number of complete movements performed during one minute.
Movement Frequency- Chair Coordination test | week 8
  Participants will be instructed to perform antiphase movements of knee flexion and extension on an instrumented chair. Intralimb spatiotemporal parameters per cycle of successive peak extension positions, and averaged per minute will include movement frequency: the number of complete movements performed during one minute.
Workload- Chair Coordination test | Baseline
  Participants will be instructed to perform antiphase movements of knee flexion and extension on an instrumented chair. Intralimb spatiotemporal parameters per cycle of successive peak extension positions, and averaged per minute will include workload (movement frequency*movement amplitude): average amplitude multiplied by the frequency, to quantify the interaction pattern.
Workload- Chair Coordination test | Day 7
  Participants will be instructed to perform antiphase movements of knee flexion and extension on an instrumented chair. Intralimb spatiotemporal parameters per cycle of successive peak extension positions, and averaged per minute will include workload (movement frequency*movement amplitude): average amplitude multiplied by the frequency, to quantify the interaction pattern.
Workload- Chair Coordination test | week 8
  Participants will be instructed to perform antiphase movements of knee flexion and extension on an instrumented chair. Intralimb spatiotemporal parameters per cycle of successive peak extension positions, and averaged per minute will include workload (movement frequency*movement amplitude): average amplitude multiplied by the frequency, to quantify the interaction pattern.
Motor fatigability during the 6 minutes condition | Baseline
  Motor fatigability during the 6 minutes condition (amplitude; frequency; workload): the percentage decline from the last minute (min 6) to the first minute will be calculated, based on the Distance Walking Index formula, for every coordination outcome.
Motor fatigability during the 6 minutes condition | Day 7
  Motor fatigability during the 6 minutes condition (amplitude; frequency; workload): the percentage decline from the last minute (min 6) to the first minute will be calculated, based on the Distance Walking Index formula, for every coordination outcome.
Motor fatigability during the 6 minutes condition | week 8
  Motor fatigability during the 6 minutes condition (amplitude; frequency; workload): the percentage decline from the last minute (min 6) to the first minute will be calculated, based on the Distance Walking Index formula, for every coordination outcome.
the paced auditory serial addition test (PASAT) | Baseline
  the paced auditory serial addition test (PASAT) to measure the cognitive fatigability
the paced auditory serial addition test (PASAT) | Day 7
  the paced auditory serial addition test (PASAT) to measure the cognitive fatigability
the paced auditory serial addition test (PASAT) | week 8
  the paced auditory serial addition test (PASAT) to measure the cognitive fatigability
the symbol digit modality test (SDMT) | Baseline
  The Symbol Digit Modalities Test (SDMT) detects cognitive impairment in less than five minutes.
the symbol digit modality test (SDMT) | Day 7
  The Symbol Digit Modalities Test (SDMT) detects cognitive impairment in less than five minutes.
the symbol digit modality test (SDMT) | week 8
  The Symbol Digit Modalities Test (SDMT) detects cognitive impairment in less than five minutes.
The 6 minute walking test | baseline
  Participants will perform the 6-minute walking test. The distance walked in each minute will be collected to calculate the Distance Walked Index (DWI) as follow: DWI = (Distance covered in the last minute - distance covered in the first minute)/distance covered in the first minute*100.
The 6 minute walking test | Day 7
  Participants will perform the 6-minute walking test. The distance walked in each minute will be collected to calculate the Distance Walked Index (DWI) as follow: DWI = (Distance covered in the last minute - distance covered in the first minute)/distance covered in the first minute*100.
The 6 minute walking test | week 8
  Participants will perform the 6-minute walking test. The distance walked in each minute will be collected to calculate the Distance Walked Index (DWI) as follow: DWI = (Distance covered in the last minute - distance covered in the first minute)/distance covered in the first minute*100.

SECONDARY OUTCOMES:
Spatiotemporal gait parameter- Cadence | Baseline
  Participants will be equipped with five portable APDM sensors (OPAL, USA, https://www.apdm.com/wearable-sensors/) to measure spatiotemporal gait parameters. Two sensors will be strapped on their ankles, two on their wrists, and one on the sternum. Cadence (number of steps per minute) will be collected throughout the walking conditions (T25FW and 6MWT) and analyzed.
Spatiotemporal gait parameter- Cadence | day 7
  Participants will be equipped with five portable APDM sensors (OPAL, USA, https://www.apdm.com/wearable-sensors/) to measure spatiotemporal gait parameters. Two sensors will be strapped on their ankles, two on their wrists, and one on the sternum. Cadence (number of steps per minute) will be collected throughout the walking conditions (T25FW and 6MWT) and analyzed.
Spatiotemporal gait parameter- Cadence | week 8
  Participants will be equipped with five portable APDM sensors (OPAL, USA, https://www.apdm.com/wearable-sensors/) to measure spatiotemporal gait parameters. Two sensors will be strapped on their ankles, two on their wrists, and one on the sternum. Cadence (number of steps per minute) will be collected throughout the walking conditions (T25FW and 6MWT) and analyzed.
Spatiotemporal gait parameter- Stride length | Baseline
  Participants will be equipped with five portable APDM sensors (OPAL, USA, https://www.apdm.com/wearable-sensors/) to measure spatiotemporal gait parameters. Two sensors will be strapped on their ankles, two on their wrists, and one on the sternum. Stride length (anteroposterior distance between two consecutive heel contact of the same foot, in meters) will be collected throughout the walking conditions (T25FW and 6MWT) and analyzed.
Spatiotemporal gait parameter- Stride length | Day 7
  Participants will be equipped with five portable APDM sensors (OPAL, USA, https://www.apdm.com/wearable-sensors/) to measure spatiotemporal gait parameters. Two sensors will be strapped on their ankles, two on their wrists, and one on the sternum. Stride length (anteroposterior distance between two consecutive heel contact of the same foot, in meters) will be collected throughout the walking conditions (T25FW and 6MWT) and analyzed.
Spatiotemporal gait parameter- Stride length | week 8
  Participants will be equipped with five portable APDM sensors (OPAL, USA, https://www.apdm.com/wearable-sensors/) to measure spatiotemporal gait parameters. Two sensors will be strapped on their ankles, two on their wrists, and one on the sternum. Stride length (anteroposterior distance between two consecutive heel contact of the same foot, in meters) will be collected throughout the walking conditions (T25FW and 6MWT) and analyzed.
Spatiotemporal gait parameter- Gait speed | Baseline
  Participants will be equipped with five portable APDM sensors (OPAL, USA, https://www.apdm.com/wearable-sensors/) to measure spatiotemporal gait parameters. Two sensors will be strapped on their ankles, two on their wrists, and one on the sternum. Gait Speed (distance divided by time- meters per second) will be collected throughout the walking conditions (T25FW and 6MWT) and analyzed.
Spatiotemporal gait parameter- Gait speed | Day 7
  Participants will be equipped with five portable APDM sensors (OPAL, USA, https://www.apdm.com/wearable-sensors/) to measure spatiotemporal gait parameters. Two sensors will be strapped on their ankles, two on their wrists, and one on the sternum. Gait Speed (distance divided by time- meters per second) will be collected throughout the walking conditions (T25FW and 6MWT) and analyzed.
Spatiotemporal gait parameter- Gait speed | week 8
  Participants will be equipped with five portable APDM sensors (OPAL, USA, https://www.apdm.com/wearable-sensors/) to measure spatiotemporal gait parameters. Two sensors will be strapped on their ankles, two on their wrists, and one on the sternum. Gait Speed (distance divided by time- meters per second) will be collected throughout the walking conditions (T25FW and 6MWT) and analyzed.
Spatiotemporal gait parameter- Double support | Baseline
  Participants will be equipped with five portable APDM sensors (OPAL, USA, https://www.apdm.com/wearable-sensors/) to measure spatiotemporal gait parameters. Two sensors will be strapped on their ankles, two on their wrists, and one on the sternum. Double Support (relative values related to the gait cycle, in percentage, that both feet are in contact with the ground) will be collected throughout the walking conditions (T25FW and 6MWT) and analyzed.
Spatiotemporal gait parameter- Double support | Day 7
  Participants will be equipped with five portable APDM sensors (OPAL, USA, https://www.apdm.com/wearable-sensors/) to measure spatiotemporal gait parameters. Two sensors will be strapped on their ankles, two on their wrists, and one on the sternum. Double Support (relative values related to the gait cycle, in percentage, that both feet are in contact with the ground) will be collected throughout the walking conditions (T25FW and 6MWT) and analyzed.
Spatiotemporal gait parameter- Double support | week 8
  Participants will be equipped with five portable APDM sensors (OPAL, USA, https://www.apdm.com/wearable-sensors/) to measure spatiotemporal gait parameters. Two sensors will be strapped on their ankles, two on their wrists, and one on the sternum. Double Support (relative values related to the gait cycle, in percentage, that both feet are in contact with the ground) will be collected throughout the walking conditions (T25FW and 6MWT) and analyzed.
Short Form of the International Physical Activity Questionnaire (IPAQ-SF) | Baseline
  Physical activity questionnaire, the short form contains 9-items and records the activity of four intensity levels: 1) vigorous-intensity activity such as aerobics, 2) moderate-intensity activity such as leisure cycling, 3) walking, and 4) sitting.
Short Form of the International Physical Activity Questionnaire (IPAQ-SF) | Day 7
  Physical activity questionnaire, the short form contains 9-items and records the activity of four intensity levels: 1) vigorous-intensity activity such as aerobics, 2) moderate-intensity activity such as leisure cycling, 3) walking, and 4) sitting.
Short Form of the International Physical Activity Questionnaire (IPAQ-SF) | week 8
  Physical activity questionnaire, the short form contains 9-items and records the activity of four intensity levels: 1) vigorous-intensity activity such as aerobics, 2) moderate-intensity activity such as leisure cycling, 3) walking, and 4) sitting.
Physical activity by means of step count | Baseline
  the participants will be asked to use the accelerometer (Actigraph) during 5 days in a roll.
Physical activity by means of step count | day 7
  the participants will be asked to use the accelerometer (Actigraph) during 5 days in a roll.
Physical activity by means of step count | week 8
  the participants will be asked to use the accelerometer (Actigraph) during 5 days in a roll.
the MFIS (modified fatigue impact scale) | Baseline
  The Modified fatigue impact scale is a 21-item questionnaire, questioning the impact of fatigue, and self-reported trait of fatigue, where higher values indicate more fatigue (maximum score of 84 points) and lower values (minimum score of 0) means less fatigue.
the MFIS (modified fatigue impact scale) | Day 7
  The Modified fatigue impact scale is a 21-item questionnaire, questioning the impact of fatigue, and self-reported trait of fatigue, where higher values indicate more fatigue (maximum score of 84 points) and lower values (minimum score of 0) means less fatigue.
the MFIS (modified fatigue impact scale) | week 8
  The Modified fatigue impact scale is a 21-item questionnaire, questioning the impact of fatigue, and self-reported trait of fatigue, where higher values indicate more fatigue (maximum score of 84 points) and lower values (minimum score of 0) means less fatigue.
The Pittsburgh Sleep Quality Index (PSQI) | baseline
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire that assesses sleep quality and disturbances over a 1-month time interval. The component scores are summed to produce a global score (range from 0 to 21). Higher scores indicate worse sleep quality and lower scores better sleep quality.
The Pittsburgh Sleep Quality Index (PSQI) | Day 7
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire that assesses sleep quality and disturbances over a 1-month time interval. The component scores are summed to produce a global score (range from 0 to 21). Higher scores indicate worse sleep quality and lower scores better sleep quality.
The Pittsburgh Sleep Quality Index (PSQI) | week 8
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire that assesses sleep quality and disturbances over a 1-month time interval. The component scores are summed to produce a global score (range from 0 to 21). Higher scores indicate worse sleep quality and lower scores better sleep quality.
Multiple Sclerosis Walking Scale-12 item (MSWS-12) | baseline
  The Multiple Sclerosis Walking Scale-12 item (MSWS-12) is a self-reported scale with to identify how people with multiple sclerosis perceived their walking ability. The questionnaire has 12 questions, with a minimum sum of 12 points and a maximum of 60 points. After, these values are transformed into a scale with a range from 0 to 100. Higher scores indicate a greater impact on walking than lower scores.
Multiple Sclerosis Walking Scale-12 item (MSWS-12) | Day 7
  The Multiple Sclerosis Walking Scale-12 item (MSWS-12) is a self-reported scale with to identify how people with multiple sclerosis perceived their walking ability. The questionnaire has 12 questions, with a minimum sum of 12 points and a maximum of 60 points. After, these values are transformed into a scale with a range from 0 to 100. Higher scores indicate a greater impact on walking than lower scores.
Multiple Sclerosis Walking Scale-12 item (MSWS-12) | week 8
  The Multiple Sclerosis Walking Scale-12 item (MSWS-12) is a self-reported scale with to identify how people with multiple sclerosis perceived their walking ability. The questionnaire has 12 questions, with a minimum sum of 12 points and a maximum of 60 points. After, these values are transformed into a scale with a range from 0 to 100. Higher scores indicate a greater impact on walking than lower scores.
25-foot walk test (T25FW) | Baseline
  Walk as fast as possible in 7.62 meters corridor
25-foot walk test (T25FW) | Day 7
  Walk as fast as possible in 7.62 meters corridor
25-foot walk test (T25FW) | week 8
  Walk as fast as possible in 7.62 meters corridor
the nine-hole peg test (NHPT) | Baseline
  Measure of manual dexterity for both hands
the nine-hole peg test (NHPT) | Day 7
  Measure of manual dexterity for both hands
the nine-hole peg test (NHPT) | week 8
  Measure of manual dexterity for both hands
the 6-minute walking test | Baseline
  Distance travelled in every minute and total distance travelled during 6 minute walking
the 6-minute walking test | Day 7
  Distance travelled in every minute and total distance travelled during 6 minute walking
the 6-minute walking test | week 8
  Distance travelled in every minute and total distance travelled during 6 minute walking
VAS (visual analogue scale) | Baseline
  The Visual Analogue Scale (VAS), will access the perceived fatigue during the 6-minute walking test, and the seated interlimb coordination test. The VAS will be asked every minute. The VAS range from 0 (no fatigue) to 10 (extremely fatigued).
VAS (visual analogue scale) | Day 7
  The Visual Analogue Scale (VAS), will access the perceived fatigue during the 6-minute walking test, and the seated interlimb coordination test. The VAS will be asked every minute. The VAS range from 0 (no fatigue) to 10 (extremely fatigued).
VAS (visual analogue scale) | week 8
  The Visual Analogue Scale (VAS), will access the perceived fatigue during the 6-minute walking test, and the seated interlimb coordination test. The VAS will be asked every minute. The VAS range from 0 (no fatigue) to 10 (extremely fatigued).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Feys, prof. dr., Principal Investigator — Hasselt University; Cintia Ramari Ferreira, dr., Study Director — Hasselt University
Locations (2):
- Belgium (2):
  - Noorderhart Revalidatie & MS centrum, Overpelt
  - National MS Center Melsbroek, Overpelt

REFERENCES:
- [Derived] Santinelli FB, Ramari C, Poncelet M, Severijns D, Kos D, Pau M, Kalron A, Meyns P, Feys P. Between-Day Reliability of the Gait Characteristics and Their Changes During the 6-Minute Walking Test in People With Multiple Sclerosis. Neurorehabil Neural Repair. 2024 Feb;38(2):75-86. doi: 10.1177/15459683231222412. Epub 2024 Jan 16. PMID 38229519